CLINICAL TRIAL: NCT04201834
Title: Risperidone for the Treatment of Huntington's Disease Chorea
Brief Title: Risperidone for the Treatment of Huntington's Disease Involuntary Movements
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ruth Schneider, MD, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4443
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Huntington Disease; Chorea
MeSH Terms: conditions — Huntington Disease; Chorea | interventions — Risperidone

STUDY DESIGN:
Masking Description: Outcomes assessor will be masked to the visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Risperidone (Experimental): Participants will initiate risperidone 0.5 mg nightly the day after the baseline visit. Dose assessment will occur at pre-specified intervals during the titration phase (week 2, 3, 4, 6, 7). The investigator will increase the dose by 0.5 mg at the week 2, week 3, week 4, and week 6 visits until either optimal chorea benefit has been obtained, an intolerable adverse event occurs, or the maximum allowable dose (3.0 mg) is reached.
  Interventions: Drug: Risperidone; Device: BioStamp nPoint device

INTERVENTIONS:
Drug: Risperidone — capsule or tablet, 0.5 mg
Device: BioStamp nPoint device — MC10 has developed the BioStamp nPointTM, a FDA 510(k) cleared medical device. This multimodal, reusable and rechargeable biosensor uses flexible and stretchable electronics to enable unobtrusive wear on the body and monitoring in the home. The sensors have accelerometry, gyroscopy, and ECG/EMG capabilities. A docking station enables wireless recharging and data collection.

SUMMARY:
The purpose of this study is to assess the safety and benefit of risperidone for the treatment of chorea (involuntary movements) in Huntington's disease. Risperidone is commonly used in clinical practice to treat chorea, however, it has not been approved by the Food and Drug Administration (FDA) to treat chorea. This study will examine 1) whether the investigators see MRI changes with risperidone treatment and 2) whether sensors applied to the participants body can measure chorea and detect changes in chorea.

ELIGIBILITY:
Inclusion Criteria:

* Manifest HD (Diagnostic Confidence Level 4 + CAG repeat ≥ 37 or family history of HD)
* UHDRS Total Maximal Chorea (TMC) ≥ 8
* UHDRS Total Functional Capacity ≥ 5
* Subject willing and able to provide written informed consent OR legally authorized representative provides written informed consent and subject provides assent*
* Between 18 and 65 years of age

Exclusion Criteria:

* Use of antipsychotic, levodopa, dopamine agonist, monoamine oxidase inhibitor or other disallowed medication in the 30 days prior to the baseline visit (see Section 4.2.5)*
* Prior non-response to risperidone or intolerability to risperidone (in the investigator's opinion)
* Allergy or hypersensitivity to risperidone
* Dysphagia that in the investigator's opinion would preclude participation in the study
* Active suicidal ideation or psychiatric condition that in the investigator's opinion would preclude study participation
* QTc > 460 msec for women and QTc > 450 msec for men on 12-lead EKG
* History of cardiac arrhythmia or congenital long QT syndrome
* Significant renal impairment (creatinine clearance < 30 mL/min as estimated by the Cockgroft-Gault formula) or hepatic impairment (AST or ALT > 2.5 times upper limit of normal OR alkaline phosphatase or total bilirubin > 2 times upper limit of normal)
* Active drug or alcohol abuse or dependence
* Pregnant or breast-feeding
* Any contraindication to MRI (e.g. pacemakers, aneurysm clips, metallic prostheses, shrapnel fragments, claustrophobia)
* History of active (clinically significant) skin disorder that would interfere with sensor adherence
* History of allergic response to adhesives
* Pacemaker, AICD, or other implantable stimulator
* Use of an investigational drug in the 30 days prior to the baseline visit
* Inability to complete study activities, as determined by the study team
* Clinically significant parkinsonism as determined by expert investigator assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- URMC Neurology; 919 Westfall Rd, Building C, Suite 100, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Risperidone
Started | 6
Completed | 5
Not Completed | 1
Not completed — Screen fail | 1

BASELINE CHARACTERISTICS:
Arm/Group | Risperidone
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Unified Huntington's Disease (HD) Rating Scale Total Maximal Chorea (UHDRS TMC) Score
Description: The UHDRS is a validated assessment of HD. The TMC score is a subset of the overall motor assessment and measures maximal chorea in seven different body regions. The TMC score ranges from 0 to 28 with higher scores indicating more chorea.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | -2.4 [-7.6 to 2.8]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.27, Paired T-Test

2. Secondary Outcome: Change From Baseline in Mean Unified Huntington's Disease (HD) Rating Scale Total Motor Score
Description: The UHDRS total motor score measures motor function. The score ranges from 0-124 . Higher total scores indicate worse motor function.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | -.02 [-5.5 to 5.1]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.92, Paired T-Test

3. Secondary Outcome: Change From Baseline in Mean Epworth Sleepiness Scale (ESS)
Description: This tool measures excessive daytime sleepiness with higher scores indicating worse health outcomes. The scale range is 0 to 24.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | 1.2 [-2.0 to 4.4]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.36, Paired T-Test

4. Secondary Outcome: Change From Baseline in Mean Barnes Akathisia Scale Global Clinical Assessment of Akathisia Item Score
Description: This tool measures drug-induced akathisia by objective observation and subjective questions. The Global Clinical Assessment of Akathisia Item score ranges from 0 to 5 with higher scores indicating more severe akathisia.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | -0.2 [-1.2 to 0.8]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.62, Paired T-Test

5. Secondary Outcome: Number of Participants With a Change in Clinical Global Impression of Change (CGI)
Description: This tool is a observer-rated scale that measures impression of severity and change. It is rated on a 7 point scale from 1(very much improved) to 7 (very much worse).
Time Frame: Baseline to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Risperidone
Number analyzed (Participants) | 5
Participants
  Minimally Improved | 3
  No Change | 1
  Minimally Worse | 1

6. Secondary Outcome: Number of Participants With a Change in Patient Global Impression of Change (PGI)
Description: This tool is a patient related scale that measures impression of change on a 7 point scale from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline to week 12
Population: PGI data were missing for one participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Risperidone
Number analyzed (Participants) | 4
Participants
  Minimally Improved | 3
  Minimally Worse | 1

7. Secondary Outcome: Change From Baseline in Mean Quantitative Motor (Q-Motor) Right Hand Speeded Finger Tapping Variability
Description: The Q-motor tool uses force transducers and a grip device to measure chorea completing four different tasks that assess fine motor finger and foot tapping speed, pronation/supination and gripping strength. With finger tapping inter-onset interval variability, which is measured in seconds, lower values indicate less irregularity and higher values more irregularity.
Time Frame: Baseline to week 8
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Risperidone
Number analyzed (Participants) | 5
seconds | -0.04 [-0.09 to 0.01]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.11, Paired T-Test

8. Secondary Outcome: Change From Baseline in Mean Short Problem Behavior Assessment (Short PBA-S) Irritability and Aggression Score
Description: This tool measures different behavioral problems which are rated for both severity and frequency on a 5 point scale; severity and frequency ratings are then multiplied to provide an overall score for each symptom. The range for the composite Irritability and Aggression score is 0-32. Higher scores indicate greater difficulties.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | 3.4 [0.8 to 6.0]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.02, Paired T-Test

9. Secondary Outcome: Columbia Suicide Severity Rating Scale( C-SSRS)
Description: The number of participants expressing suicidal ideations will be determined by answering yes to any of the following questions: Have you wished you were dead or wished you could go to sleep and not wake up?, Have you actually had any thoughts of killing yourself?, Have you been thinking about how you might do this?, Have you had these thoughts and had some intention of acting on them?, Have you started to work out or worked out the details of how to kill yourself? Do you intend to carry out this plan? All questions require only a yes or no response. There is no numerical scoring or rating.
Time Frame: Baseline to week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Risperidone
Number analyzed (Participants) | 5
Participants
  Suicidal Ideation - Yes | 0
  Suicidal Ideation - No | 5

10. Secondary Outcome: Change From Baseline in Mean Apathy Scale Score
Description: This tool measures the presence and severity of apathy. The range is 0 to 42 with higher scores indicating worse health outcomes
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | 0.8 [-11.4 to 12.9]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.86, Paired T-Test

11. Secondary Outcome: Change From Baseline in Mean Hospital Anxiety and Depression Scale-Depression Score
Description: This is a self-reported scale that measures anxiety and depression. The Depression sub-score ranges from 0 to 21 with higher scores indicating more depressive symptoms.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | -1.0 [-3.2 to 1.2]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.27, Paired T-Test

12. Secondary Outcome: Change From Baseline in Mean Montreal Cognitive Assessment
Description: The Montreal Cognitive assessment (MoCA) measures cognitive function (attention and concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation). The score ranges from 0 to 30. Lower scores indicate worse cognitive function.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | -0.6 [-3.6 to 2.4]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.61, Paired T-Test

13. Secondary Outcome: Change From Baseline in Mean Unified Huntington's Disease (HD) Rating Scale Independence Scale Score
Description: The UHDRS Independence Scale measures level of current functional independence. The score ranges from 10 to 100 with higher scores indicating a higher degree of functional independence.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | 4.0 [-7.1 to 15.1]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.37, Paired T-Test

14. Secondary Outcome: Change From Baseline in Mean Hospital Anxiety and Depression Scale-Anxiety Score
Description: This is a self-reported scale that measures anxiety and depression. The Anxiety sub-score ranges from 0 to 21 with higher scores indicating more anxiety symptoms.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone
Number analyzed (Participants) | 5
score on a scale | -1.4 [-4.6 to 1.8]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.30, Paired T-Test

15. Secondary Outcome: Change From Baseline in MC10-Assessed Mean Gait Cadence
Description: MC10 BioStamp nPoint is a wearable biosensor system with accelerometry, gyroscopy, and ECG/EMG capabilities that provides various gait metrics. Gait cadence refers to steps per minute. Higher values indicate more steps per minute.
Time Frame: Screening to Week 8
Population: Sensor data were missing for one participant.
Measure: Mean (95% Confidence Interval); unit: steps per minute
Arm/Group | Risperidone
Number analyzed (Participants) | 4
steps per minute | 0.6 [-7.5 to 8.8]
Statistical Analysis 1: Comparison: Risperidone; Test type: Superiority; p = 0.82, Paired t-test

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Our definitions of adverse events and serious adverse events is consistence with the definitions that are provided by clinicaltrials.gov. The recording of adverse events began once the participant signed informed consent and continued until the participant completed the study or withdrew from participation.
Arm/Group | Risperidone
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Risperidone (N=5)
Prolonged QTc Interval (Cardiac disorders) | 1
Tics (Congenital, familial and genetic disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Hyperemia (Injury, poisoning and procedural complications) | 1
Somnolence (Nervous system disorders) | 1
Anxiety (Nervous system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Constant throat clearing (Nervous system disorders) | 1
Jerky movements - hands, arms, shoulders (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT04201834/Prot_SAP_001.pdf